CLINICAL TRIAL: NCT05053724
Title: Efficacy of the "Start to Move" Protocol on Functionality, Delirium and Acquired Weakness in ICU. Randomized Clinical Trial.
Brief Title: Efficacy of the "Start to Move" Protocol on Functionality, Delirium and Acquired Weakness in ICU
Acronym: STM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Felix Bulnes (Other)
Responsible Party: Principal Investigator, Sebastian Soto López, Physical Therapist, Hospital Felix Bulnes
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: starttomove
Record Dates: First submitted 2021-05-28; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Intensive Care Unit Acquired Weakness; Intensive Care Unit Delirium; Intensive Care Neuropathy; Intensive Care Unit Syndrome; Mechanical Ventilation Complication
Keywords: Intensive Care Unit; Early mobilization; Physical therapy; ICU acquired weakness; Funcionality; Invasive mechanical ventilation

STUDY DESIGN:
Intervention Model Description: Methods: Randomized, single-blind, controlled clinical trial. Computational random assignment of the intervention using sealed envelopes (1:1), non-probabilistic, consecutive sampling of subjects admitted to Clínica Ensenada ICU between January 2018 - July 2019 and who met selection criteria.
  Participants: All subjects admitted to Clínica Ensenada ICU, adults ≥15 years with invasive mechanical ventilation requirement >48 hours were recruited. Subjects with neuromuscular disease; psychiatric history (attempted autolysis, schizophrenia, senile dementia or others, who due to their condition are not able to follow a logical sequential order, which could bias the evaluation and functional treatment); limb amputation; pregnancy; cardiorespiratory arrest with severe hypoxic-ischemic brain damage; total dependence prior to hospitalization, according to Barthel index (<20 points); and not consenting to participate in the study were excluded.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study was conducted in a single 12-bed ICU clinical center, during 2018-2019. Subjects who met the inclusion criteria were asked for informed consent from the responsible guardian and were subsequently randomized (1:1) into Start to move group and conventional treatment group. Sequentially numbered sealed envelopes were used for allocation, which were accessed only by research personnel not participating in the clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start to move group (Experimental): In the Start to move group, physical therapy was included according to the Gosselink protocol, which establishes 6 levels of care divided according to system stability and state of consciousness. At level 0, no physical mobilization therapy was applied due to systemic lability. From level 1 to 5, passive mobilizations, use of muscle electrostimulation, active mobilizations and exercises against resistance, application of conventional cycloergometer, up to walking with assistance if the subject is able to perform it.
  Interventions: Other: Star to move Protocol
- Conventional treatment group (Active Comparator): In the conventional treatment group, passive mobilization, active-assisted mobilization and exercises against resistance, facilitation of high functional positions such as sedentary, bipedal and walking were applied, according to conventional treatment protocol.
  Interventions: Other: Star to move Protocol

INTERVENTIONS:
Other: Star to move Protocol — Progressive physical therapy according to the Gosslink protocol called "Start to move".

SUMMARY:
Background: ICU hospitalization is associated with loss of strength, functionality and delirium. The "Start to Move protocol" demonstrated efficacy in improving and minimizing such effects.

Aim: To evaluate the effectiveness of the "Start to move protocol" compared with conventional treatment in ICU subjects on functionality, weakness acquired in the Intensive Care Unit (ICU-AW), incidence of delirium, days of invasive mechanical ventilation (IMV), ICU stay and 28-day mortality.

Methods: Randomized controlled clinical trial. Including adults ≥15 years with IMV >48 hours, randomized into Start to move and conventional treatment groups.Functionality, ICU-AW incidence, delirium incidence, IMV days, ICU stay and mortality-28 days were analyzed.

DETAILED DESCRIPTION:
Introduction:

Individuals hospitalized in Intensive Care Units are subjected to a prolonged state of rest and to various factors that directly or indirectly affect the muscular and organic structure, which can result in ICU-acquired weakness (ICU-AW) and a limitation in functional performance.

These factors can be divided into metabolic, pharmacological and organic, where sustained hyperglycemia, corticosteroid use, sedation-analgesia, neuromuscular blockade and multiorgan failure associated with sepsis or septic shock stand out. This state translates into a direct loss of muscle mass, specifically of type II fibers, physiologically explained by an increase in the myosin protein degradation process, a decrease in protein synthesis and an increase in proinflammatory cells that favor the weakness of the critically ill patient.

Brower et al. studied that the effects of prolonged rest produce a deconditioning and atrophy of the musculature. After 14 days of immobilization, young people and adults are exposed to a 9% loss of quadriceps muscle mass, which translates into a loss of muscle strength of up to 27%.In subjects subjected to invasive mechanical ventilation, it has been shown that the cross-sectional area of the quadriceps muscle can decrease up to 12.5% in the first week of their stay in the ICU, which can increase up to 15.7% if they present multiorgan failure versus a 3% loss in subjects with single organ failure.

ICU-AW and loss of function are also directly related to the prolonged use of sedoanalgesia, neuromuscular blockade and a higher incidence of delirium in the ICU. The presence of delirium is related to low participation in physical therapies, either by decreased cooperation and/or psychomotor agitation, thus directly influencing muscle status and subsequent functional recovery.

Brummel et al. report that delirium is common in the ICU, affecting between 60-80% of subjects undergoing IMV and between 20-50% of subjects on noninvasive mechanical ventilation, increasing the risk of removal of invasive elements, accidental extubations and the need for physical restraints that may delay the onset of functional recovery.

To demonstrate the consequences of prolonged rest and quantify ICU-AW, the Medical Research Council (MRC) assessment scale is used, a validated tool which analytically measures the strength of six muscle groups bilaterally with a score of 30 points per hemibody, obtaining a total of 60 points. A score of 48 points or less determines the presence of ICU-AW.

On the other hand, the validated Functional Status Scale - Intensive Care Unit (FSS-ICU), which measures functional milestones with a score between 0 and 35 points, is commonly used to assess the functionality of the critically ill patient 12.

The aim of our study is to evaluate the effectiveness of the Start to move protocol compared to conventional ICU treatment on functionality, ICU-Aw, incidence of delirium, days of mechanical ventilation, ICU stay and 28-day mortality, Clínica Ensenada 2018 - 2019.

ELIGIBILITY:
Inclusion Criteria:

* Subjects admitted to ICU
* Adults ≥15 years
* IMV requirement >48 hours

Exclusion Criteria:

* Neuromuscular disease
* Psychiatric history (attempted autolysis, schizophrenia, senile dementia or others, who due to their condition are unable to follow simple orders, which could bias the assessment and functional treatment)
* Limb amputation
* Pregnancy
* Cardiorespiratory arrest with severe hypoxic-ischemic brain damage
* Total dependence prior to hospitalization, according to Barthel index (<20 points);
* Subject without consenting to participate in the study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Change of ICU-acquired weakness | It is measured in the first 24 hours of the awakening phase of the patient in the 24 hours prior to discharge from the ICU.
  ICU-AW was measured through the MRC scale of 60 points, where scores below 48 points indicate ICU-AW and more than 48 points the greater the strength of the subject.
Change of Functionality of the Critically Ill Patient (Intra-hospital) | It is measured in the first 24 hours of the awakening phase of the patient in the 24 hours prior to discharge from the ICU.
  Through the FSS-ICU evaluation scale, a score of 0 to 35 points is made to evaluate the motor function of the critical patient, where the higher the score, the greater the subject's functionality.
Change of Functionality of the Critically Ill Patient (pre-hospitalization) | It is measured in the first 24 hours of the awakening phase of the patient in the 24 hours prior to discharge from the ICU.
  Evaluation of the Barthel index of a family member, of the baseline state of the patient, before hospitalization. The total score is 100 points, the higher the score, the better the patient's baseline functionality.
Change of Delirium | It is measured in the first 24 hours of the awakening phase of the patient in the 24 hours prior to discharge from the ICU.
  It is measured using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) scale to determine the presence of delirium. It does not have a score, if it meets criteria the subject will have delirium.

SECONDARY OUTCOMES:
ICU stay (days) | It is measured in the 24 hours prior to discharge from the ICU.
  Number of days hospitalized in ICU, up to 45 days. From the date of admission to the ICU until the departure from the ICU.
Days of invasive mechanical ventilation (IMV) | It is measured in the 24 hours prior to discharge from the ICU.
  Number of days of invasive mechanical ventilation during hospitalization, up to 45 days. From the day of intubation until weaning from invasive mechanical ventilation.
Mortality at 28 days, post ICU discharge | Measured at 28 days post ICU discharge.
  The patient's death is verified according to the medical record (during hospitalization) or through a telephone number to a family member (outside the hospital).

CONTACTS AND LOCATIONS:
Locations (1):
- Sebastián Eduardo Soto López, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
Data were recorded using an Epidata form.

REFERENCES:
- [Result] Schefold JC, Bierbrauer J, Weber-Carstens S. Intensive care unit-acquired weakness (ICUAW) and muscle wasting in critically ill patients with severe sepsis and septic shock. J Cachexia Sarcopenia Muscle. 2010 Dec;1(2):147-157. doi: 10.1007/s13539-010-0010-6. Epub 2010 Dec 17. PMID 21475702
- [Result] Nordon-Craft A, Moss M, Quan D, Schenkman M. Intensive care unit-acquired weakness: implications for physical therapist management. Phys Ther. 2012 Dec;92(12):1494-506. doi: 10.2522/ptj.20110117. Epub 2012 Jan 26. PMID 22282769
- [Result] Sommers J, Engelbert RH, Dettling-Ihnenfeldt D, Gosselink R, Spronk PE, Nollet F, van der Schaaf M. Physiotherapy in the intensive care unit: an evidence-based, expert driven, practical statement and rehabilitation recommendations. Clin Rehabil. 2015 Nov;29(11):1051-63. doi: 10.1177/0269215514567156. Epub 2015 Feb 13. PMID 25681407
- [Result] Brower RG. Consequences of bed rest. Crit Care Med. 2009 Oct;37(10 Suppl):S422-8. doi: 10.1097/CCM.0b013e3181b6e30a. PMID 20046130
- [Result] Suetta C, Hvid LG, Justesen L, Christensen U, Neergaard K, Simonsen L, Ortenblad N, Magnusson SP, Kjaer M, Aagaard P. Effects of aging on human skeletal muscle after immobilization and retraining. J Appl Physiol (1985). 2009 Oct;107(4):1172-80. doi: 10.1152/japplphysiol.00290.2009. Epub 2009 Aug 6. PMID 19661454
- [Result] Jones SW, Hill RJ, Krasney PA, O'Conner B, Peirce N, Greenhaff PL. Disuse atrophy and exercise rehabilitation in humans profoundly affects the expression of genes associated with the regulation of skeletal muscle mass. FASEB J. 2004 Jun;18(9):1025-7. doi: 10.1096/fj.03-1228fje. Epub 2004 Apr 14. PMID 15084522
- [Result] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Result] Kamdar BB, Combs MP, Colantuoni E, King LM, Niessen T, Neufeld KJ, Collop NA, Needham DM. The association of sleep quality, delirium, and sedation status with daily participation in physical therapy in the ICU. Crit Care. 2016 Aug 18;19:261. doi: 10.1186/s13054-016-1433-z. PMID 27538536
- [Result] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527
- [Result] Thrush A, Rozek M, Dekerlegand JL. The clinical utility of the functional status score for the intensive care unit (FSS-ICU) at a long-term acute care hospital: a prospective cohort study. Phys Ther. 2012 Dec;92(12):1536-45. doi: 10.2522/ptj.20110412. Epub 2012 Sep 6. PMID 22956427
- [Result] de Jonghe B, Lacherade JC, Sharshar T, Outin H. Intensive care unit-acquired weakness: risk factors and prevention. Crit Care Med. 2009 Oct;37(10 Suppl):S309-15. doi: 10.1097/CCM.0b013e3181b6e64c. PMID 20046115
- [Result] Kho ME, Truong AD, Zanni JM, Ciesla ND, Brower RG, Palmer JB, Needham DM. Neuromuscular electrical stimulation in mechanically ventilated patients: a randomized, sham-controlled pilot trial with blinded outcome assessment. J Crit Care. 2015 Feb;30(1):32-9. doi: 10.1016/j.jcrc.2014.09.014. Epub 2014 Sep 22. PMID 25307979
- [Result] Parry SM, Berney S, Koopman R, Bryant A, El-Ansary D, Puthucheary Z, Hart N, Warrillow S, Denehy L. Early rehabilitation in critical care (eRiCC): functional electrical stimulation with cycling protocol for a randomised controlled trial. BMJ Open. 2012 Sep 13;2(5):e001891. doi: 10.1136/bmjopen-2012-001891. Print 2012. PMID 22983782
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Schweickert WD, Pohlman MC, Pohlman AS, Nigos C, Pawlik AJ, Esbrook CL, Spears L, Miller M, Franczyk M, Deprizio D, Schmidt GA, Bowman A, Barr R, McCallister KE, Hall JB, Kress JP. Early physical and occupational therapy in mechanically ventilated, critically ill patients: a randomised controlled trial. Lancet. 2009 May 30;373(9678):1874-82. doi: 10.1016/S0140-6736(09)60658-9. Epub 2009 May 14. PMID 19446324
- [Derived] Soto S, Adasme R, Vivanco P, Figueroa P. Efficacy of the "Start to move" protocol on functionality, ICU-acquired weakness and delirium: A randomized clinical trial. Med Intensiva (Engl Ed). 2024 Apr;48(4):211-219. doi: 10.1016/j.medine.2024.01.003. Epub 2024 Feb 23. PMID 38402053